CLINICAL TRIAL: NCT03091036
Title: Impact of a Proactive and Integrated Health Intervention Between Different Assistance Levels Over Some Indicators in the Care of Chronic Complex Patient (CCP)
Brief Title: Impact of a Health Intervention on Some Indicators in the Care of Chronic Complex Patient (CCP).
Acronym: CCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: María José del Olmo Rubio (Other)
Collaborators: Hospital Universitario 12 de Octubre (Other)
Responsible Party: Sponsor-Investigator, María José del Olmo Rubio, Principal investigator, Hospital Universitario 12 de Octubre
Organization: Hospital Universitario 12 de Octubre (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: InveCuidPCC16
Record Dates: First submitted 2017-03-16; First posted 2017-03-27 (Actual); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Preventive Care
Keywords: Chronic; Complex
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Proactive healthcare intervention (Other): Participants who were included before (single-arm pre-post study), now a proactive and integrated intervention program for the health is performed of the complex chronic patient, based in an improvement of the care process.
  Interventions: Other: Proactive healthcare intervention

INTERVENTIONS:
Other: Proactive healthcare intervention — There is an intervention in the coordination of health resources, and monitoring readmissions and know the benefit in total cost of care in 4 month.

SUMMARY:
The aim of this study is to assess the effectiveness of proactive and integrated healthcare program for chronic complex patients (CCP). This program are based in coordination the primary level of attention with and speciality level. The objective is reducing hospital readmissions and know the benefit in total cost of care in 4 month before and 4 after intervention.

DETAILED DESCRIPTION:
Quasi-experimental study with single-arm (pre-post study design without control group). The investigators checking pre and post intervention the effectiveness of a healthcare program for CCP. The interventions consist:

1. - Help the nurse in the hospital to carry out the care plans and the continuity care report.
2. - Refer patients to the social workers.
3. - Collaborate with the social worker to refer to centers of media, long stay and reference hospital.
4. - Ensure the follow-up appointments for the CCP.
5. - Make proactive calls to the CCP and/or their caregiver after discharge
6. - Plan the hospital discharge 48 hours in advance, so that the family and the patient can be organized.

The investigator analysed if with this program, the CCP reducing hospital readmission and reducing the Hospital expenditure.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 75 years.
* Having attended 5 or more emergency visits or having had more than 3 hospital admissions in the last 12 months.
* Identified with social risk alert.

Exclusion Criteria:

* Participate in other health programs (AHT, diabetes mellitus,...).
* Terminal patient.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Pre-post change in days of Hospital stay from baseline to 16 weeks. | Baseline and 16 weeks.
  The same group of patients are analyzed the days of hospital stay at the end of 16 weeks of follow-up pre intervention (baseline) and 16 week after the intervention.

SECONDARY OUTCOMES:
Number of hospital readmissions visits for CCP change from baseline to 16 weeks. | Baseline and 16 weeks.
  The same group of patients are analyzed the number of hospital readmissions visit for CCP at the end of 16 weeks pre intervention (considered baseline) of follow-up and 16 weeks after the intervention.
Number of urgency visits for CCP change from baseline to 16 weeks. | Baseline and 16 weeks.
  The same group of patients are analyzed the number of urgency visits and primary care visit for CCP at the end of 16 weeks pre intervention (considered baseline) of follow-up and 16 weeks after the intervention.
Number of primary care visits for CCP change from baseline to 16 weeks. | Baseline and 16 weeks.
  The same group of patients are analyzed the number of primary care visits for CCP at the end of 16 weeks pre intervention (considered baseline) of follow-up and 16 weeks after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: María José del Olmo Rubio, Principal Investigator — Hospital 12 de Octubre de Madrid
Locations (1):
- Hospital Universitario 12 de Octubre de Madrid, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No